CLINICAL TRIAL: NCT00259506
Title: Implementation and Evaluation of "Mindfulness-Based Cognitive Therapy" in a Health Care Region in Flanders: a Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Ministry of the Flemish Community (Other Government)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2005/195
Record Dates: First submitted 2005-11-28; First posted 2005-11-29 (Estimated); Last update posted 2009-06-03 (Estimated); Status verified 2009-06

CONDITIONS: Recurrent Depression
Keywords: Recurrent depression; Mental Health
MeSH Terms: conditions — Depression; Psychological Well-Being | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Mindfulness-Based Cognitive Therapy (MBCT)

SUMMARY:
Research project regarding the possibility to implement and the efficacy of a non-drug, psychotherapeutic intervention (MBCT), in preventing relapse/recurrence of depression.

DETAILED DESCRIPTION:
This trial is based on the following publications:

Teasdale JD, Segal ZV, Williams JMG, Ridgeway VA, Soulsby JM, Lau MA. Prevention of relapse / recurrence in major depression by Mindfulness-Based Cognitive Therapy. Journal of Consulting and Clinical Psychology 2000; 68(4): 615-623.

Ma SH, Teasdale JD. Mindfulness-Based Cognitive Therapy for depression: replication and exploration of differential relapse prevention effects. Journal of Consulting and Clinical Psychology 2004; 72(1): 31-40.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years and above
* place of residence in accordance with a well-defined region (pilot study)
* given informed consent
* diagnosis of recurrent depression (DSM-IV-TR)
* at least 3 depressive episodes in the anamnesis (depression: either primary or secondary diagnosis)
* last depressive episode at least 8 weeks ago (DSM-IV-TR)
* absence of a present depressive episode
* history of treatment by an antidepressant medication
* HRSD-score <14 at baseline assessment (Hamilton Rating Scale for Depression, HRSD-17)
* absence of exclusion criteria

Exclusion Criteria:

* based on DSM-IV-TR: current diagnosis of any of the following psychiatric disorders: lifetime mood disorder, chronic depression, dysthymia, current substance abuse, obsessive-compulsive disorder, bipolar disorder, acute psychosis, cognitive disorder, organic mental disorder, pervasive developmental disorder, mental retardation, primary diagnosis of axis-II-disorder, at risk for suicide
* Extended experience with zen- or vipassana meditation (or mindfulness) in the past or
* more than 1 hour practice of zen- or vipassana meditation (or mindfulness) per week during the last 8 weeks
* other meditation practices except for MBCT during the training
* more than 1 psychiatric consultation per 3-4 weeks during the training and follow-up
* intensive psychotherapy during the training and follow-up
* schizophrenia or schizoaffective disorder in the anamnesis
* physical problems which make it difficult to participate in the programme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Estimated)
Dates: Start 2006-03; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Feasibility to implement MBCT in a Flemish region
Relapse/recurrence of depression after approximately 12 months

SECONDARY OUTCOMES:
Health status
Quality of life
Coping
Fear
Rumination

CONTACTS AND LOCATIONS:
Overall Officials: Kees van Heeringen, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be